CLINICAL TRIAL: NCT06209242
Title: Cast Immobilization Versus Percutaneous Pinning in Local Anesthesia for Extra-articular Fracture of Distal End Radius in an Elderly Patient: a Prospective Randomized Controlled Study
Brief Title: Cast Immobilization Versus Percutaneous Pinning for Fracture of Radius in an Elderly Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 027/2564
Record Dates: First submitted 2023-12-20; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Closed Fracture of Lower End of Radius

STUDY DESIGN:
Intervention Model Description: This prospective randomized controlled trial enrolled participants aged over 60 years with AO23-A2 or AO23-A3 distal radius fractures and no contraindications for local anesthesia. The participants were randomly assigned to either the cast immobilization or percutaneous pinning group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cast immobilization (Experimental): Using cast immobilization with sugar tong and short arm splinting
  Interventions: Procedure: Cast immobilization
- Percutaneous pinning (Experimental): Using k-wire percutaneous pinning
  Interventions: Procedure: Percutaneous pinning

INTERVENTIONS:
Procedure: Percutaneous pinning — Using k- wire percutaneous pinning with local anesthesia with one-day surgery protocol
  Arms: Percutaneous pinning
Procedure: Cast immobilization — Using sugar tong slab and then replace to short arm casting within 1 week
  Arms: Cast immobilization

SUMMARY:
Distal radius fractures, particularly in elderly individuals, are a common problem associated with increasing age and hormonal changes. The choice of treatment, such as cast immobilization or percutaneous pinning, plays a crucial role in achieving optimal functional outcomes and facilitating a return to normal activities. This study aimed to compare the radiological and clinical outcomes of cast immobilization and percutaneous pinning in elderly patients with distal radius fractures.

DETAILED DESCRIPTION:
Background: Distal radius fractures, particularly in elderly individuals, are a common problem associated with increasing age and hormonal changes. The choice of treatment, such as cast immobilization or percutaneous pinning, plays a crucial role in achieving optimal functional outcomes and facilitating a return to normal activities. This study aimed to compare the radiological and clinical outcomes of cast immobilization and percutaneous pinning in elderly patients with distal radius fractures.

Methods: This prospective randomized controlled trial enrolled participants aged over 60 years with AO23-A2 or AO23-A3 distal radius fractures and no contraindications for local anesthesia. The participants were randomly assigned to either the cast immobilization or percutaneous pinning group. Follow-up was conducted for 3 months, during which radiological outcomes and clinical outcomes were assessed. Radiological parameters included radial angulation, while clinical outcomes were evaluated using the Disability of Arm, Shoulder, and Hand (DASH) score, range of motion, and grip strength. Additionally, data on complications and pain levels measured using the Visual Analog Scale (VAS) were collected for the percutaneous pinning group under local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* aged >60 years
* primary distal end radius fracture type AO23-A2 or AO23-A3

Exclusion Criteria:

* multiple trauma
* onset > 2 weeks
* systemic diseases such as RA
* steroid user
* contraindication for LA

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Radiological parameters | 1 wk , 4 wk , 3 months
  Radial angulation, radial inclination, ulnar deviation, radial height

SECONDARY OUTCOMES:
DASH score | 1 month, 3 months
  Functional outcome
Hand function | 1 month, 3 months
  Range of motion, grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Teerasit Punprasitwech, MD, Principal Investigator — QSMVH
Locations (1):
- Queen Savang Vadhana Memorial hospital, Chon Buri, Sriracha, Thailand

IPD SHARING:
Plan to Share IPD: No
Data was save inform of excel, sheets and SPSS